CLINICAL TRIAL: NCT01798836
Title: Oestradiol Pre-treatment in an Ultrashort Flare GnRH Agonist/GnRH Antagonist Protocol in Poor Responders Undergoing IVF
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Obtained results were not good. Protocol was proved ineffective.
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Assistant Professor in Obstetrics and Gynecology/Assisted Reproduction, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030675
Record Dates: First submitted 2013-02-20; First posted 2013-02-26 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: IVF/ICSI cycles, poor responders, ultrashort flare protocol, antagonist protocol
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oestradiol and ultrashort GnRH agonist/antagonist protocol (Experimental): Women will begin pretreatment with 4 mg/day of 17 β-estradiol before the combination of GnRH ultashort agonist and antagonist protocol
  Interventions: Procedure: Oestradiol pre-treatment and combination of GnRH agonist/antagonist protocol
- GnRH agonist or antagonist protocol. (Active Comparator): Women will undergo either a conventional short or long GnRH agonist or an antagonist protocol during COH for IVF
  Interventions: Procedure: GnRH agonist or antagonist protocol without oestradiol pre-treatment

INTERVENTIONS:
Procedure: Oestradiol pre-treatment and combination of GnRH agonist/antagonist protocol
  Arms: Oestradiol and ultrashort GnRH agonist/antagonist protocol
Procedure: GnRH agonist or antagonist protocol without oestradiol pre-treatment
  Arms: GnRH agonist or antagonist protocol.

SUMMARY:
To evaluate the effect of oestradiol pre-treatment in a combined ultrashort flare GnRH agonist /GnRH antagonist protocol

DETAILED DESCRIPTION:
The combined ultrashort flare GnRH agonist /GnRH antagonist protocol during COH cycle resulted in a significantly higher clinical pregnancy rate in patients with poor embryo quality, with repeated IVF failures and in poor responders. This is a protocol combining the effect of the microdose flare on endogenous FSH release with the benefit of an immediate LH suppression of the GnRH antagonist.

A major disadvantage of the use of a GnRH antagonist protocol is the limitation for programming cycles, as the drugs administration is started on day 2 of the menstrual cycle and is strictly followed until the hCG criteria are met.

The purpose of the study is to perform oestradiol pre-treatment with the combined ultrashort flare GnRH agonist /GnRH antagonist protocol aiming to

1. better programme an antagonist cycle and
2. improve the IVF outcome parameters, from the production of more follicles / oocytes up to the rise in live birth rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with poor or no response in previous COH for IVF cycles
* Patients with AMH < 1 and/or FSH >12
* Poor quality of embryos in previous cycles
* Age of patients up to 44 years

Exclusion Criteria:

* Patients with normal ovarian reserve
* Patients with sonographically detected hydrosalpinges
* Presence of intramural fibroid distorting the endometrial cavity or submucous myoma or Asherman's syndrome
* Women with thrombofilia disorders

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 2 years
Clinical pregnancy rate | 2 years

SECONDARY OUTCOMES:
Number of oocytes retrieved | 2 years
Top embryo quality at day 2 | 2 years
Biochemical pregnancy | 2 years
Ectopic pregnancy | 2 years
Miscarriage rate | 2 years

OTHER OUTCOMES:
Positive Pregnancy Test | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George Salamalekis, MD, PhD, Principal Investigator — National and Kapodistrian University of Athens; Charalampos Siristatidis, Assistant Professor, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Assisted Reproduction Unit, 3rd Department of Obstetrics and Gynecology. Attikon University Hospital, Athens, Attica, Greece

REFERENCES:
- [Background] Griesinger G, Kolibianakis EM, Venetis C, Diedrich K, Tarlatzis B. Oral contraceptive pretreatment significantly reduces ongoing pregnancy likelihood in gonadotropin-releasing hormone antagonist cycles: an updated meta-analysis. Fertil Steril. 2010 Nov;94(6):2382-4. doi: 10.1016/j.fertnstert.2010.04.025. Epub 2010 May 26. PMID 20537631
- [Background] Bosch E. Can we skip weekends in GnRH antagonist cycles without compromising the final outcome? Fertil Steril. 2012 Jun;97(6):1299-300. doi: 10.1016/j.fertnstert.2012.04.024. No abstract available. PMID 22656307
- [Result] Orvieto R, Nahum R, Rabinson J, Gemer O, Anteby EY, Meltcer S. Ultrashort flare GnRH agonist combined with flexible multidose GnRH antagonist for patients with repeated IVF failures and poor embryo quality. Fertil Steril. 2009 Apr;91(4 Suppl):1398-400. doi: 10.1016/j.fertnstert.2008.04.064. Epub 2008 Aug 3. PMID 18675974
- [Result] Cedrin-Durnerin I, Guivarc'h-Leveque A, Hugues JN; Groupe d'Etude en Medecine et Endocrinologie de la Reproduction. Pretreatment with estrogen does not affect IVF-ICSI cycle outcome compared with no pretreatment in GnRH antagonist protocol: a prospective randomized trial. Fertil Steril. 2012 Jun;97(6):1359-64.e1. doi: 10.1016/j.fertnstert.2012.02.028. Epub 2012 Mar 28. PMID 22464760